CLINICAL TRIAL: NCT00537238
Title: A Randomized, Double-Blind, Parallel-Group Multi-Center Comparative Flexible-Dose Study Of Pregabalin Versus Levetiracetam As Adjunctive Therapy To Reduce Seizure Frequency In Subjects With Partial Seizures
Brief Title: Pregabalin Versus Levetiracetam In Partial Seizures
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: A0081157
Record Dates: First submitted 2007-09-27; First posted 2007-10-01 (Estimated); Results first posted 2013-07-11 (Estimated); Last update posted 2021-01-28 (Actual); Status verified 2013-05

CONDITIONS: Partial Seizures
Keywords: Epilepsies partial; Partial Seizure Disorder; Complex Partial Seizure Disorder; Epilepsy
MeSH Terms: conditions — Seizures; Epilepsies, Partial; Epilepsy, Complex Partial; Epilepsy | interventions — Pregabalin; Levetiracetam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- B (Active Comparator)
  Interventions: Drug: pregabalin
- A (Active Comparator)
  Interventions: Drug: levetiracetam

INTERVENTIONS:
Drug: pregabalin — 300, 450, 600 mg/day administered orally, BID until seizure control/improvement or intolerable side effects
  Arms: B
Drug: levetiracetam — 1000, 2000, 3000 mg/day administered orally, BID until seizure control/improvement or intolerable side effects
  Arms: A

SUMMARY:
This study will compare pregabalin and levetiracetam in patients with partial seizures. It will also evaluate the safety and tolerability of pregabalin and levetiracetam in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Subjects (male or female) must be > 18 years of age, with a diagnosis of epilepsy with partial seizures, as defined in the International League Against Epilepsy (ILAE) classification of seizures.
* Partial seizures may be simple or complex, with or without secondary tonic-clonic generalization.
* Subjects must be have been diagnosed with epilepsy for at least 2 years, and must have been unresponsive to treatment with at least two but no more than five prior antiepileptic drugs (AEDs), and at the time of study enrollment are on stable dosages of 1 or 2 standard AEDs.

Exclusion Criteria:

* Females who are pregnant, breastfeeding, or intend to become pregnant during the course of the trial will be excluded
* Subjects with other neurologic illness that could impair endpoint assessment, or subjects with Lennox-Gastaut syndrome, absence seizures, status epileptics within the 12 months prior to trial entry, or with seizures due to an underlying medical illness or metabolic syndrome, will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 509 (Actual)
Dates: Start 2007-10; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (62):
- Belgium (2):
  - Pfizer Investigational Site, Duffel
  - Pfizer Investigational Site, Yvoir
- Bulgaria (5):
  - Pfizer Investigational Site, Kyustendil
  - Pfizer Investigational Site, Pernik
  - Pfizer Investigational Site, Plovdiv
  - Pfizer Investigational Site, Rousse
  - Pfizer Investigational Site, Sofia
- Colombia (2):
  - Pfizer Investigational Site, Barranquilla, Atlántico
  - Pfizer Investigational Site, Bogota, Cundinamarca
- Costa Rica (2):
  - Pfizer Investigational Site, Montes de Oca, Provincia de San José
  - Pfizer Investigational Site, San José
- Czechia (7):
  - Pfizer Investigational Site, Brno
  - Pfizer Investigational Site, Hradec Králové
  - Pfizer Investigational Site, Olomouc
  - Pfizer Investigational Site, Ostrava-Trebovice
  - Pfizer Investigational Site, Prague
  - Pfizer Investigational Site, Příbram
  - Pfizer Investigational Site, Rychnov nad Kněžnou
- France (2):
  - Pfizer Investigational Site, Strasbourg
  - Pfizer Investigational Site, Toulouse
- Germany (2):
  - Pfizer Investigational Site, Bonn
  - Pfizer Investigational Site, Hamburg
- Greece (2):
  - Pfizer Investigational Site, Athens
  - Pfizer Investigational Site, Thessaloniki
- India (3):
  - Pfizer Investigational Site, Pune, Maharashtra
  - Pfizer Investigational Site, Chandigarh, Punjab
  - Pfizer Investigational Site, Ludhiana, Punjab
- Italy (4):
  - Pfizer Investigational Site, Florence
  - Pfizer Investigational Site, Foggia
  - Pfizer Investigational Site, Pisa
  - Pfizer Investigational Site, Siena
- Lithuania (2):
  - Pfizer Investigational Site, Kaunas
  - Pfizer Investigational Site, Vilnius
- Mexico (2):
  - Pfizer Investigational Site, Distrito Federal
  - Pfizer Investigational Site, San Luis Potosí City
- Pfizer Investigational Site, Panama City, Panama
- Pfizer Investigational Site, Lima, Peru
- Philippines (6):
  - Pfizer Investigational Site, Tondo, Manila
  - Pfizer Investigational Site, Cebu City
  - Pfizer Investigational Site, Davao City
  - Pfizer Investigational Site, Makati City
  - Pfizer Investigational Site, Manila
  - Pfizer Investigational Site, Quezon City
- Russia (2):
  - Pfizer Investigational Site, Moscow
  - Pfizer Investigational Site, Saint Petersburg
- South Korea (3):
  - Pfizer Investigational Site, Busan
  - Pfizer Investigational Site, Daejeon
  - Pfizer Investigational Site, Seoul
- Spain (6):
  - Pfizer Investigational Site, Donostia / San Sebastian, Guipuzcoa
  - Pfizer Investigational Site, Alicante
  - Pfizer Investigational Site, Barcelona
  - Pfizer Investigational Site, Córdoba
  - Pfizer Investigational Site, Girona
  - Pfizer Investigational Site, Seville
- Taiwan (3):
  - Pfizer Investigational Site, Kaohsiung City
  - Pfizer Investigational Site, Taichung
  - Pfizer Investigational Site, Tainan
- Turkey (Türkiye) (3):
  - Pfizer Investigational Site, Çapa, Istanbul
  - Pfizer Investigational Site, Ankara
  - Pfizer Investigational Site, Cerrahpasa / Istanbul
- Venezuela (2):
  - Pfizer Investigational Site, Caracas, Libertador
  - Pfizer Investigational Site, Caracas, Miranda

REFERENCES:
- [Derived] Zaccara G, Almas M, Pitman V, Knapp L, Posner H. Efficacy and safety of pregabalin versus levetiracetam as adjunctive therapy in patients with partial seizures: a randomized, double-blind, noninferiority trial. Epilepsia. 2014 Jul;55(7):1048-57. doi: 10.1111/epi.12679. Epub 2014 Jun 5. PMID 24902473

RESULTS

PARTICIPANT FLOW:
Groups:
- Pregabalin: Pregabalin 75 milligram (mg) capsule orally twice daily (BID) for 1 Week followed by pregabalin 150 mg orally BID up to Week 4 in the titration phase (TP). If seizure control was inadequate (adequate: at least [>=] 50% reduction in seizures), pregabalin dose was escalated to 225 mg orally BID for Week 2 through Week 4. Participants who had adequate seizure control with pregabalin 150 mg or 225 mg orally BID dose in TP, continued same dose during the 12-week maintenance phase(MP). Participants who had inadequate seizure control, received pregabalin 300 mg orally BID during MP. Participants also received placebo matched to levetiracetam capsule orally BID along with pregabalin during TP and MP. After MP, participants were allowed to progress into optional (opt) blinded continuation phase, and remained on dose from MP for a maximum of 2 years or until last participant either completed or discontinued from MP. Participants underwent an end-of-study medication taper over a 1-week period.
- Levetiracetam: Levetiracetam 500 mg capsule orally BID for 2 Weeks in the TP. If seizure control was inadequate (adequate: >= 50% reduction in seizures), the levetiracetam dose was escalated to 1000 mg orally BID for Week 2 through Week 4. Participants who had adequate seizure control with levetiracetam 500 or 1000 mg orally BID dose in the TP, continued same dose in the 12-week MP. Participants who had inadequate seizure control, received levetiracetam 1500 mg orally BID during the MP. Participants also received placebo matched to pregabalin capsule orally BID along with levetiracetam during TP and MP. After the MP, participants were allowed to progress into the opt blinded continuation phase, and remained on the dose from the MP for a maximum of 2 years or until the last participant either completed or discontinued from the MP. Participants underwent an end-of-study medication taper over a 1-week period.
Period: Overall Study
Arm/Group | Pregabalin | Levetiracetam
Started | 254 | 255
Completed Titration Phase | 226 | 236
Completed Maintenance Phase | 208 (Primary analysis drawn from the population in the maintenance phase.) | 210 (Primary analysis drawn from the population in the maintenance phase.)
Entered Opt Blinded Continuation Phase | 185 (Participants who had clinical benefit were eligible to progress into opt blinded continuation phase.) | 195 (Participants who had clinical benefit were eligible to progress into opt blinded continuation phase.)
Completed | 80 (Completed designates participants who completed the opt blinded continuation phase.) | 82 (Completed designates participants who completed the opt blinded continuation phase.)
Not Completed | 174 | 173
Not completed — Death | 1 | 2
Not completed — Adverse Event | 31 | 22
Not completed — Lack of Efficacy | 20 | 21
Not completed — Lost to Follow-up | 12 | 8
Not completed — Withdrawal by Subject | 51 | 47
Not completed — Protocol Violation | 15 | 19
Not completed — Does not meet entrance criteria | 0 | 2
Not completed — Other | 44 | 52

BASELINE CHARACTERISTICS:
Groups:
- Pregabalin: Pregabalin 75 mg capsule orally BID for 1 Week followed by pregabalin 150 mg orally BID up to Week 4 in the TP. If seizure control was inadequate (adequate: >=50% reduction in seizures), the pregabalin dose was escalated to 225 mg orally BID for Week 2 through 4. Participants who had adequate seizure control with pregabalin 150 mg or 225 mg orally BID dose in TP, continued same dose during the 12-week MP. Participants who had inadequate seizure control, received pregabalin 300 mg orally BID during the MP. Participants also received placebo matched to levetiracetam capsule orally BID along with pregabalin during the TP and the MP. After the MP, participants were allowed to progress into the opt blinded continuation phase, and remained on dose from the MP for a maximum of 2 years or until the last participant either completed or discontinued from MP. Participants underwent an end-of-study medication taper over a 1-week period.
- Total: Total of all reporting groups
Arm/Group | Pregabalin | Levetiracetam | Total
Number analyzed (Participants) | 254 | 255 | 509
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.7 (11.2) | 36.3 (12.2) | 34.5 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 134 | 130 | 264
  Male | 120 | 125 | 245

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants With Response to Treatment
Description: Participants who had at least 50% reduction in 28-day seizure rate from baseline to the end of the maintenance phase were considered as responders. The 28-day seizure rate was calculated as number of partial seizures in the period divided by difference of number of days in the period and number of missing diary day entries in the period, multiplied by 28.
Time Frame: Baseline up to Week 16
Population: Per protocol population included all randomized participants who had at least 28 days of study drug during the maintenance phase and a minimum of 28 days of utilizable seizure diary data during baseline and maintenance phases of the study and had no major protocol violation.
Measure: Number; unit: proportion of participants
Arm/Group | Pregabalin | Levetiracetam
Number analyzed (Participants) | 164 | 177
proportion of participants | 0.59 | 0.59
Statistical Analysis 1: Comparison: Pregabalin vs Levetiracetam; Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the difference in proportion (Pregabalin - Levetiracetam) was greater than -0.12; Difference in Proportion = 0.00, 90% CI 2-sided [-0.08 to 0.09]

2. Secondary Outcome: Percent Change From Baseline in 28 Day Seizure Frequency at Week 16
Description: The seizures were recorded by the participants, by a family member, by a caregiver, or by a legal guardian and documented in a daily seizure diary. Participant's 28-day seizure frequency of all partial seizure was assessed during double blind (TP + MP) phase compared with baseline.
Time Frame: Baseline, Week 16
Population: Full analysis set (FAS) included all randomized participants who had received at least 1 blinded dose of study drug and had at least 1 baseline and post baseline primary efficacy evaluation.
Measure: Median (Full Range); unit: percent change
Arm/Group | Pregabalin | Levetiracetam
Number analyzed (Participants) | 253 | 254
percent change | -53.93 [-100.0 to 533.1] | -57.28 [-100.0 to 276.9]
Statistical Analysis 1: Comparison: Pregabalin vs Levetiracetam; Rank analysis of covariance (ANCOVA) model was used to derive p-value with treatment as main effect and cluster as cofactor, percent change in 28-day seizure counts between baseline and treatment periods as dependent variable. Median differences and 95% confidence interval (CI) were based on Hodges-Lehmann estimation; Test type: Superiority or Other; p = 0.3571, Ranked ANCOVA; Median difference = 4.1, 95% CI 2-sided [-2.6 to 10.9]

3. Secondary Outcome: Change From Baseline in the Proportion of 28-day Secondarily Generalized Tonic-clonic (SGTC) Seizure Rate to 28-day All Partial Seizure Rate at Week 16
Description: Change was calculated as (proportion of SGTC seizure rate divided by all partial seizure rates during double blind phase) minus (proportion of SGTC seizure rate divided by all partial seizure rates at baseline). Negative values indicated reductions in seizures.
Time Frame: Baseline, Week 16
Population: SGTC population included all participants who had at least 1 SGTC seizure during either baseline or double-blind phase. n=number of participants evaluable at specific time points for each arm group, respectively.
Measure: Mean (Standard Deviation); unit: percentage of all partial seizure/28days
Arm/Group | Pregabalin | Levetiracetam
Number analyzed (Participants) | 107 | 111
percentage of all partial seizure/28days
  Baseline (n=107, 111) | 39.41 (38.141) | 38.94 (35.870)
  Change at Week 16 (n=102, 101) | 3.93 (30.158) | 6.33 (32.071)

4. Secondary Outcome: Percentage of Participants Without Seizures
Description: Seizure free for 28 days was defined as participants who have not experienced any seizure (simple partial, complex partial and SGTC) for at least 28 consecutive days from their last seizure until the end of the maintenance phase. Same participant could be seizure free for a specific type of seizure but not necessarily for the other types of seizure.
Time Frame: Baseline up to Week 16
Population: FAS included all randomized participants who had received at least 1 blinded dose of study drug and had at least 1 baseline and post baseline primary efficacy evaluation. N (number of participants analyzed)=participants who were evaluable for this measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pregabalin | Levetiracetam
Number analyzed (Participants) | 201 | 210
percentage of participants
  All Partial Seizure | 19.9 [14.4 to 25.4] | 27.6 [21.6 to 33.7]
  Simple Partial Seizure | 65.7 [59.1 to 72.2] | 66.2 [59.8 to 72.6]
  Complex Partial Seizure | 49.3 [42.3 to 56.2] | 59.0 [52.4 to 65.7]
  SGTC Seizure | 80.6 [75.1 to 86.1] | 79.0 [73.5 to 84.6]
Statistical Analysis 1: Comparison: Pregabalin vs Levetiracetam; All partial seizure: p-value was calculated from the 2-sided Fisher's exact test; Test type: Superiority or Other; p = 0.0822, Fisher Exact
Statistical Analysis 2: Comparison: Pregabalin vs Levetiracetam; Simple partial seizure: p-value was calculated from the 2-sided Fisher's exact test; Test type: Superiority or Other; p = 0.9175, Fisher Exact
Statistical Analysis 3: Comparison: Pregabalin vs Levetiracetam; Complex partial seizure: p-value was calculated from the 2-sided Fisher's exact test; Test type: Superiority or Other; p = 0.0483, Fisher Exact
Statistical Analysis 4: Comparison: Pregabalin vs Levetiracetam; SGTC seizure: p-value was calculated from the 2-sided Fisher's exact test; Test type: Superiority or Other; p = 0.7139, Fisher Exact

5. Secondary Outcome: Change From Baseline in Brief Psychiatric Rating Scale - Anchored (BPRS-A) Total and Core Score at Week 7, 10, 13, 16 and Follow-up
Description: BPRS-A:18-item clinician rated scale assesses somatic concern,anxiety, emotional withdrawal,conceptual disorganization,hallucinatory behavior(HB), guilt feelings,suspiciousness,disorientation,tension,mannerisms and posturing,grandiosity,depressive mood,hostility,motor retardation,uncooperativeness,unusual thought content,blunted affect,excitement. Items rated on 7-point scale 1 (not reported) to 7 (very severe). Total score=sum of items(range 18-126), core score=sum of conceptual disorganization, suspiciousness, HB, unusual thought content(range 4-28). Higher total/core score=more impairment.
Time Frame: Baseline, Week 7, 10, 13, 16 and Follow-up (Day 7 of taper phase)
Population: FAS included all randomized participants who had received at least 1 blinded dose of study drug and had at least 1 baseline and post baseline primary efficacy evaluation. n=number of participants evaluable at specific time points for each arm group, respectively.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Pregabalin | Levetiracetam
Number analyzed (Participants) | 253 | 254
units on a scale
  Baseline: Total BPRS-A Score (n=253, 254) | 27.26 (0.55) | 26.09 (0.56)
  Baseline: Core BPRS-A Score (n=253, 254) | 5.18 (0.13) | 5.01 (0.13)
  Change at Week 7: Total BPRS-A Score (n=217, 225) | -2.16 (0.36) | -1.70 (0.36)
  Change at Week 7: Core BPRS-A Score (n=216, 225) | -0.34 (0.08) | -0.22 (0.08)
  Change at Week 10: Total BPRS-A Score (n=217, 219) | -2.64 (0.37) | -2.42 (0.38)
  Change at Week 10: Core BPRS-A Score (n=217, 219) | -0.40 (0.08) | -0.34 (0.08)
  Change at Week 13: Total BPRS-A Score (n=209, 214) | -2.99 (0.39) | -2.68 (0.39)
  Change at Week 13: Core BPRS-A Score (n=209, 214) | -0.51 (0.07) | -0.38 (0.07)
  Change at Week 16: Total BPRS-A Score (n=235, 241) | -2.70 (0.40) | -1.92 (0.40)
  Change at Week 16: Core BPRS-A Score (n=235, 241) | -0.40 (0.08) | -0.26 (0.08)
  Change at Follow-up: Total BPRS-A Score(n=178,189) | -2.77 (0.44) | -1.42 (0.43)
  Change at Follow-up: Core BPRS-A Score(n=178,189) | -0.37 (0.10) | -0.11 (0.10)
Statistical Analysis 1: Comparison: Pregabalin vs Levetiracetam; Baseline, total BPRS score: ANCOVA model was used to calculate LS mean estimates of the treatment difference along with 95% CI, with main effects of treatment and combined center, and for post-baseline assessments baseline was included as a covariate; Test type: Superiority or Other; p = 0.1334, ANCOVA; Least squares (LS) mean difference = 1.17, 95% CI 2-sided [-0.36 to 2.69], Standard Error of Mean 0.78
Statistical Analysis 2: Comparison: Pregabalin vs Levetiracetam; Baseline, core BPRS score: ANCOVA model was used to calculate LS mean estimates of the treatment difference along with 95% CI, with main effects of treatment and combined center, and for post-baseline assessments baseline was included as a covariate; Test type: Superiority or Other; p = 0.3551, ANCOVA; LS mean differences = 0.17, 95% CI 2-sided [-0.19 to 0.52], Standard Error of Mean 0.18
Statistical Analysis 3: Comparison: Pregabalin vs Levetiracetam; Change at Week 7, total BPRS score: ANCOVA model was used to calculate LS mean estimates of the treatment difference along with 95% CI, with main effects of treatment and combined center, and for post-baseline assessments baseline was included as a covariate; Test type: Superiority or Other; p = 0.3638, ANCOVA; LS mean differences = -0.46, 95% CI 2-sided [-1.45 to 0.53], Standard Error of Mean 0.50
Statistical Analysis 4: Comparison: Pregabalin vs Levetiracetam; Change at Week 7, core BPRS score: ANCOVA model was used to calculate LS mean estimates of the treatment difference along with 95% CI, with main effects of treatment and combined center, and for post-baseline assessments baseline was included as a covariate; Test type: Superiority or Other; p = 0.2457, ANCOVA; LS mean differences = -0.12, 95% CI 2-sided [-0.34 to 0.09], Standard Error of Mean 0.11
Statistical Analysis 5: Comparison: Pregabalin vs Levetiracetam; Change at Week 10, total BPRS score: ANCOVA model was used to calculate LS mean estimates of the treatment difference along with 95% CI, with main effects of treatment and combined center, and for post-baseline assessments baseline was included as a covariate; Test type: Superiority or Other; p = 0.6640, ANCOVA; LS mean differences = -0.23, 95% CI 2-sided [-1.26 to 0.81], Standard Error of Mean 0.53
Statistical Analysis 6: Comparison: Pregabalin vs Levetiracetam; Change at Week 10, core BPRS score: ANCOVA model was used to calculate LS mean estimates of the treatment difference along with 95% CI, with main effects of treatment and combined center, and for post-baseline assessments baseline was included as a covariate; Test type: Superiority or Other; p = 0.5950, ANCOVA; LS mean differences = -0.06, 95% CI 2-sided [-0.30 to 0.17], Standard Error of Mean 0.12
Statistical Analysis 7: Comparison: Pregabalin vs Levetiracetam; Change at Week 13, total BPRS score: ANCOVA model was used to calculate LS mean estimates of the treatment difference along with 95% CI, with main effects of treatment and combined center, and for post-baseline assessments baseline was included as a covariate; Test type: Superiority or Other; p = 0.5701, ANCOVA; LS mean differences = -0.31, 95% CI 2-sided [-1.38 to 0.76], Standard Error of Mean 0.55
Statistical Analysis 8: Comparison: Pregabalin vs Levetiracetam; Change at Week 13, core BPRS score: ANCOVA model was used to calculate LS mean estimates of the treatment difference along with 95% CI, with main effects of treatment and combined center, and for post-baseline assessments baseline was included as a covariate; Test type: Superiority or Other; p = 0.2452, ANCOVA; LS mean differences = -0.12, 95% CI 2-sided [-0.33 to 0.08], Standard Error of Mean 0.10
Statistical Analysis 9: Comparison: Pregabalin vs Levetiracetam; Change at Week 16, total BPRS score: ANCOVA model was used to calculate LS mean estimates of the treatment difference along with 95% CI, with main effects of treatment and combined center, and for post-baseline assessments baseline was included as a covariate; Test type: Superiority or Other; p = 0.1697, ANCOVA; LS mean differences = -0.77, 95% CI 2-sided [-1.88 to 0.33], Standard Error of Mean 0.56
Statistical Analysis 10: Comparison: Pregabalin vs Levetiracetam; Change at Week 16, core BPRS score: ANCOVA model was used to calculate LS mean estimates of the treatment difference along with 95% CI, with main effects of treatment and combined center, and for post-baseline assessments baseline was included as a covariate; Test type: Superiority or Other; p = 0.2283, ANCOVA; LS mean differences = -0.14, 95% CI 2-sided [-0.36 to 0.09], Standard Error of Mean 0.11
Statistical Analysis 11: Comparison: Pregabalin vs Levetiracetam; Change at Follow-up, total BPRS score: ANCOVA model was used to calculate LS mean estimates of the treatment difference along with 95% CI, with main effects of treatment and combined center, and for post-baseline assessments baseline was included as a covariate; Test type: Superiority or Other; p = 0.0262, ANCOVA; LS mean differences = -1.35, 95% CI 2-sided [-2.54 to -0.16], Standard Error of Mean 0.61
Statistical Analysis 12: Comparison: Pregabalin vs Levetiracetam; Change at Follow-up, core BPRS score: ANCOVA model was used to calculate LS mean estimates of the treatment difference along with 95% CI, with main effects of treatment and combined center, and for post-baseline assessments baseline was included as a covariate; Test type: Superiority or Other; p = 0.0495, ANCOVA; LS mean differences = -0.26, 95% CI 2-sided [-0.52 to 0.00], Standard Error of Mean 0.13

6. Secondary Outcome: Hospital Anxiety and Depression Scale (HADS) Score
Description: HADS: participant rated questionnaire with 2 subscales. HADS-A assesses state of generalized anxiety (anxious mood, restlessness, anxious thoughts, panic attacks); HADS-D assesses state of lost interest and diminished pleasure response (lowering of hedonic tone). Each subscale comprised of 7 items with range 0 (no presence of anxiety or depression) to 3 (severe feeling of anxiety or depression). Total score 0 to 21 for each subscale; higher score indicates greater severity of anxiety and depression symptoms.
Time Frame: Baseline, Week 16
Population: FAS included all randomized participants who had received at least 1 blinded dose of study drug and had at least 1 baseline and post baseline primary efficacy evaluation. N (number of participants analyzed)=participants who were evaluable for this measure. n=number of participants evaluable at specific time points for each arm group, respectively.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Pregabalin | Levetiracetam
Number analyzed (Participants) | 253 | 253
units on a scale
  Baseline: HADS-A (n=253, 253) | 7.25 (0.26) | 7.34 (0.27)
  Baseline: HADS-D (n=253, 253) | 6.22 (0.25) | 6.00 (0.25)
  Week 16: HADS-A (n=228, 241) | 6.32 (0.22) | 6.06 (0.22)
  Week 16: HADS-D (n=228, 241) | 5.41 (0.22) | 5.42 (0.22)
Statistical Analysis 1: Comparison: Pregabalin vs Levetiracetam; Baseline, HADS-A: ANCOVA model was used to calculate LS mean estimates of the treatment difference along with 95% CI, with main effects of treatment and combined center, and for post-baseline assessments baseline was included as a covariate; Test type: Superiority or Other; p = 0.8084, ANCOVA; LS mean differences = -0.09, 95% CI 2-sided [-0.82 to 0.64], Standard Error of Mean 0.37
Statistical Analysis 2: Comparison: Pregabalin vs Levetiracetam; Baseline, HADS-D: ANCOVA model was used to calculate LS mean estimates of the treatment difference along with 95% CI, with main effects of treatment and combined center, and for post-baseline assessments baseline was included as a covariate; Test type: Superiority or Other; p = 0.5263, ANCOVA; LS mean differences = 0.22, 95% CI 2-sided [-0.47 to 0.91], Standard Error of Mean 0.35
Statistical Analysis 3: Comparison: Pregabalin vs Levetiracetam; Week 16, HADS-A: ANCOVA model was used to calculate LS mean estimates of the treatment difference along with 95% CI, with main effects of treatment and combined center, and for post-baseline assessments baseline was included as a covariate; Test type: Superiority or Other; p = 0.4008, ANCOVA; LS mean differences = 0.25, 95% CI 2-sided [-0.34 to 0.85], Standard Error of Mean 0.30
Statistical Analysis 4: Comparison: Pregabalin vs Levetiracetam; Week 16, HADS-D: ANCOVA model was used to calculate LS mean estimates of the treatment difference along with 95% CI, with main effects of treatment and combined center, and for post-baseline assessments baseline was included as a covariate; Test type: Superiority or Other; p = 0.9749, ANCOVA; LS mean differences = -0.01, 95% CI 2-sided [-0.61 to 0.59], Standard Error of Mean 0.30

7. Secondary Outcome: Medical Outcomes Study Sleep Scale (MOS-SS) Score
Description: Participant-rated 12-item questionnaire to assess constructs of sleep over past week; 7 subscales:sleep disturbance,snoring,awakened short of breath,sleep adequacy,somnolence (range:0-100);sleep quantity (range:0-24),optimal sleep(yes/no), and 9 item index measures of sleep disturbance provide composite scores:sleep problem summary,overall sleep problem. Except adequacy,optimal sleep and quantity, higher scores=more impairment. Scores transformed (actual raw score[RS] minus lowest possible score divided by possible RS range*100);total score range:0-100;higher score=more intensity of attribute.
Time Frame: Baseline, Week 16
Population: FAS included all randomized participants who had received at least 1 blinded dose of study medication and had at least 1 baseline and post baseline primary efficacy evaluation. n=number of participants evaluable at specific time points for each arm group, respectively.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Pregabalin | Levetiracetam
Number analyzed (Participants) | 253 | 254
units on a scale
  Baseline: Sleep Disturbance (n=253, 253) | 27.06 (1.45) | 28.10 (1.48)
  Baseline: Snoring (n=253, 254) | 30.72 (2.25) | 32.42 (2.29)
  Baseline: Awaken Short of Breath (n=253, 254) | 15.72 (1.54) | 17.26 (1.57)
  Baseline: Quantity of Sleep (n=252, 252) | 7.77 (0.10) | 7.82 (0.10)
  Baseline: Adequacy of Sleep (n=253, 254) | 62.96 (1.79) | 64.40 (1.83)
  Baseline: Somnolence (n=253, 254) | 34.85 (1.43) | 33.77 (1.45)
  Baseline: Sleep Problem Index (9) (n=253, 253) | 29.62 (1.16) | 29.49 (1.18)
  Week 16: Sleep Disturbance (n=230, 241) | 21.97 (1.16) | 23.61 (1.17)
  Week 16: Snoring (n=230, 240) | 33.77 (1.72) | 23.75 (1.73)
  Week 16: Awaken Short of Breath (n=230, 241) | 15.15 (1.48) | 14.27 (1.48)
  Week 16: Quantity of Sleep (n=230, 241) | 7.89 (0.09) | 7.75 (0.09)
  Week 16: Adequacy of Sleep (n=230, 241) | 63.46 (1.72) | 66.46 (1.73)
  Week 16: Somnolence (n=230, 241) | 31.56 (1.33) | 32.29 (1.34)
  Week 16: Sleep Problem Index (9) (n=230, 241) | 26.64 (0.95) | 26.00 (0.96)
Statistical Analysis 1: Comparison: Pregabalin vs Levetiracetam; Baseline sleep disturbance: ANCOVA model was used to calculate LS mean estimates of the treatment difference along with 95% CI, with main effects of treatment and combined center, for post-baseline assessments baseline was included as a covariate; Test type: Superiority or Other; p = 0.6161, ANCOVA; LS mean differences = -1.03, 95% CI 2-sided [-5.08 to 3.01], Standard Error of Mean 2.06
Statistical Analysis 2: Comparison: Pregabalin vs Levetiracetam; Week 16 sleep disturbance: ANCOVA model was used to calculate LS mean estimates of the treatment difference along with 95% CI, with main effects of treatment and combined center, for post-baseline assessments baseline was included as a covariate; Test type: Superiority or Other; p = 0.3154, ANCOVA; LS mean differences = -1.63, 95% CI 2-sided [-4.83 to 1.56], Standard Error of Mean 1.62
Statistical Analysis 3: Comparison: Pregabalin vs Levetiracetam; Baseline snoring: ANCOVA model was used to calculate LS mean estimates of the treatment difference along with 95% CI, with main effects of treatment and combined center, for post-baseline assessments baseline was included as a covariate; Test type: Superiority or Other; p = 0.5930, ANCOVA; LS mean differences = -1.70, 95% CI 2-sided [-7.94 to 4.54], Standard Error of Mean 3.18
Statistical Analysis 4: Comparison: Pregabalin vs Levetiracetam; Week 16 snoring: ANCOVA model was used to calculate LS mean estimates of the treatment difference along with 95% CI, with main effects of treatment and combined center, for post-baseline assessments baseline was included as a covariate; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS mean differences = 10.02, 95% CI 2-sided [5.27 to 14.76], Standard Error of Mean 2.42
Statistical Analysis 5: Comparison: Pregabalin vs Levetiracetam; Baseline awaken short of breath: ANCOVA model was used to calculate LS mean estimates of the treatment difference along with 95% CI, with main effects of treatment and combined center, for post-baseline assessments baseline was included as a covariate; Test type: Superiority or Other; p = 0.4807, ANCOVA; LS mean differences = -1.54, 95% CI 2-sided [-5.83 to 2.75], Standard Error of Mean 2.18
Statistical Analysis 6: Comparison: Pregabalin vs Levetiracetam; Week 16 awaken short of breath: ANCOVA model was used to calculate LS mean estimates of the treatment difference along with 95% CI, with main effects of treatment and combined center, for post-baseline assessments baseline was included as a covariate; Test type: Superiority or Other; p = 0.6708, ANCOVA; LS mean differences = 0.88, 95% CI 2-sided [-3.18 to 4.94], Standard Error of Mean 2.07
Statistical Analysis 7: Comparison: Pregabalin vs Levetiracetam; Baseline quantity of sleep: ANCOVA model was used to calculate LS mean estimates of the treatment difference along with 95% CI, with main effects of treatment and combined center, for post-baseline assessments baseline was included as a covariate; Test type: Superiority or Other; p = 0.7574, ANCOVA; LS mean differences = -0.04, 95% CI 2-sided [-0.32 to 0.24], Standard Error of Mean 0.14
Statistical Analysis 8: Comparison: Pregabalin vs Levetiracetam; Week 16 quantity of sleep: ANCOVA model was used to calculate LS mean estimates of the treatment difference along with 95% CI, with main effects of treatment and combined center, for post-baseline assessments baseline was included as a covariate; Test type: Superiority or Other; p = 0.2615, ANCOVA; LS mean differences = 0.14, 95% CI 2-sided [-0.10 to 0.38], Standard Error of Mean 0.12
Statistical Analysis 9: Comparison: Pregabalin vs Levetiracetam; Baseline adequacy of sleep: ANCOVA model was used to calculate LS mean estimates of the treatment difference along with 95% CI, with main effects of treatment and combined center, for post-baseline assessments baseline was included as a covariate; Test type: Superiority or Other; p = 0.5703, ANCOVA; LS mean differences = -1.44, 95% CI 2-sided [-6.42 to 3.54], Standard Error of Mean 2.53
Statistical Analysis 10: Comparison: Pregabalin vs Levetiracetam; Week 16 adequacy of sleep: ANCOVA model was used to calculate LS mean estimates of the treatment difference along with 95% CI, with main effects of treatment and combined center, for post-baseline assessments baseline was included as a covariate; Test type: Superiority or Other; p = 0.2160, ANCOVA; LS mean differences = -2.99, 95% CI 2-sided [-7.74 to 1.75], Standard Error of Mean 2.41
Statistical Analysis 11: Comparison: Pregabalin vs Levetiracetam; Baseline somnolence: ANCOVA model was used to calculate LS mean estimates of the treatment difference along with 95% CI, with main effects of treatment and combined center, for post-baseline assessments baseline was included as a covariate; Test type: Superiority or Other; p = 0.5952, ANCOVA; LS mean differences = 1.07, 95% CI 2-sided [-2.89 to 5.03], Standard Error of Mean 2.02
Statistical Analysis 12: Comparison: Pregabalin vs Levetiracetam; Week 16 somnolence: ANCOVA model was used to calculate LS mean estimates of the treatment difference along with 95% CI, with main effects of treatment and combined center, for post-baseline assessments baseline was included as a covariate; Test type: Superiority or Other; p = 0.6984, ANCOVA; LS mean differences = -0.72, 95% CI 2-sided [-4.40 to 2.95], Standard Error of Mean 1.87
Statistical Analysis 13: Comparison: Pregabalin vs Levetiracetam; Baseline sleep problem index (9): ANCOVA model was used to calculate LS mean estimates of the treatment difference along with 95% CI, with main effects of treatment and combined center, for post-baseline assessments baseline was included as a covariate; Test type: Superiority or Other; p = 0.9389, ANCOVA; LS mean differences = 0.13, 95% CI 2-sided [-3.09 to 3.34], Standard Error of Mean 1.64
Statistical Analysis 14: Comparison: Pregabalin vs Levetiracetam; Week 16 sleep problem index (9): ANCOVA model was used to calculate LS mean estimates of the treatment difference along with 95% CI, with main effects of treatment and combined center, for post-baseline assessments baseline was included as a covariate; Test type: Superiority or Other; p = 0.6344, ANCOVA; LS mean differences = 0.64, 95% CI 2-sided [-2.00 to 3.27], Standard Error of Mean 1.34

8. Secondary Outcome: Percentage of Participants With Optimal Sleep Assessed Using Medical Outcomes Study-Sleep Scale (MOS-SS) Score
Description: MOS-SS: participant-rated 12 item questionnaire to assess constructs of sleep over past week. It included 7 subscales: sleep disturbance, snoring, awakened short of breath, sleep adequacy, somnolence, sleep quantity and optimal sleep. Participants responded whether their sleep was optimal or not by choosing yes or no. Percentage of participants with optimal sleep are reported.
Time Frame: Baseline, Week 16
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | Pregabalin | Levetiracetam
Number analyzed (Participants) | 252 | 252
percentage of participants
  Baseline (n=252, 252) | 56.0 | 55.6
  Week 16 (n=230, 241) | 58.3 | 50.2
Statistical Analysis 1: Comparison: Pregabalin vs Levetiracetam; Baseline: Logistic regression model was used to estimate odds ratio and corresponding 95% CI of treatment difference, with treatment as fixed effect and for post-baseline assessments baseline was included as a covariate; Test type: Superiority or Other; p = 0.9285, Regression, Logistic; Odds Ratio (OR) = 1.016, 95% CI 2-sided [0.715 to 1.444]
Statistical Analysis 2: Comparison: Pregabalin vs Levetiracetam; Week 16: Logistic regression model was used to estimate odds ratio and corresponding 95% CI of treatment difference, with treatment as fixed effect and for post-baseline assessments baseline was included as a covariate; Test type: Superiority or Other; p = 0.0696, Regression, Logistic; Odds Ratio (OR) = 1.432, 95% CI 2-sided [0.972 to 2.110]

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Pregabalin | Levetiracetam
Serious Adverse Events (participants affected / at risk) | 24/254 | 24/255
Other Adverse Events (participants affected / at risk) | 148/254 | 127/255
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pregabalin (N=254) | Levetiracetam (N=255)
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Gastroduodenitis (Gastrointestinal disorders) | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1
Asthenia (General disorders) | 1 | 0
Drowning (General disorders) | 1 | 0
Polyp (General disorders) | 0 | 1
Abscess limb (Infections and infestations) | 1 | 0
Acute tonsillitis (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0
Bronchopneumonia (Infections and infestations) | 1 | 0
Pharyngotonsillitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Pulmonary tuberculosis (Infections and infestations) | 0 | 1
Septic shock (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Brain contusion (Injury, poisoning and procedural complications) | 0 | 1
Burns third degree (Injury, poisoning and procedural complications) | 1 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 1
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 1
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0
Intentional overdose (Injury, poisoning and procedural complications) | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0
Weight increased (Investigations) | 2 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal disorder (Musculoskeletal and connective tissue disorders) | 0 | 1
Retroperitoneal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Complex partial seizures (Nervous system disorders) | 0 | 1
Convulsion (Nervous system disorders) | 5 | 1
Dizziness (Nervous system disorders) | 1 | 0
Drug withdrawal convulsions (Nervous system disorders) | 0 | 1
Epilepsy (Nervous system disorders) | 1 | 2
Ischaemic stroke (Nervous system disorders) | 0 | 1
Postictal state (Nervous system disorders) | 0 | 1
Sedation (Nervous system disorders) | 0 | 1
Status epilepticus (Nervous system disorders) | 1 | 2
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Abortion threatened (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Aggression (Psychiatric disorders) | 0 | 2
Depressed mood (Psychiatric disorders) | 0 | 1
Personality change (Psychiatric disorders) | 0 | 1
Personality disorder (Psychiatric disorders) | 1 | 0
Somatoform disorder neurologic (Psychiatric disorders) | 1 | 0
Suicide attempt (Psychiatric disorders) | 0 | 2
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1
Ovarian cyst (Reproductive system and breast disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pregabalin (N=254) | Levetiracetam (N=255)
Nausea (Gastrointestinal disorders) | 5 | 15
Nasopharyngitis (Infections and infestations) | 24 | 19
Weight increased (Investigations) | 26 | 8
Dizziness (Nervous system disorders) | 59 | 42
Headache (Nervous system disorders) | 37 | 30
Somnolence (Nervous system disorders) | 83 | 76
Insomnia (Psychiatric disorders) | 5 | 15

LIMITATIONS AND CAVEATS:
Results for BPRS were provided as change in scores at Week 16 compared to baseline instead of absolute scores as per planned analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.